CLINICAL TRIAL: NCT00144456
Title: A Prospective, Randomized, Double-blind Study to Compare the Effect of ED-71 With That of Alfacalcidol on Fracture Incidence in Osteoporotic Patients
Brief Title: A New Active Vitamin D, ED-71 for Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ED-209JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — eldecalcitol; alfacalcidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ED-71; Drug: Alfacalcidol placebo
- 2 (Active Comparator)
  Interventions: Drug: Alfacalcidol; Drug: ED-71 placebo

INTERVENTIONS:
Drug: ED-71 — 0.75μg/day(p.o.)for 144 weeks
  Arms: 1
Drug: Alfacalcidol — 1.0μg/day(p.o.)for 144 weeks
  Arms: 2
Drug: ED-71 placebo — 0 μg/day(p.o.)for 144 weeks
  Arms: 2
Drug: Alfacalcidol placebo — 0 μg/day(p.o.)for 144 weeks
  Arms: 1

SUMMARY:
A prospective, randomized, double-blind study to compare the effect of ED-71 with that of alfacalcidol on fracture incidence

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic patients who meet any of the following condition:

  1. with at least one fragility fracture,
  2. above 70 year-old with bone mineral density below 70% young adult mean,
  3. with bone mineral density below 60% young adult mean
* Women three years or more after menopause or men

Exclusion Criteria:

* Current disorders such as primary hyperparathyroidism, Cushing's syndrome,gonadal insufficiency, poorly controlled diabetes mellitus or other causes of secondary osteoporosis
* A history or suspicion of active urolithiasis at any time
* Use of bisphosphonates in the past 12 months
* Use of medications known to affect bone in the past 2 months
* Abnormal serum calcium, urinary calcium, serum creatinine or liver function tests

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1056 (Actual)
Dates: Start 2004-09; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Incidences of vertebral fracture | throughout study

SECONDARY OUTCOMES:
Changes of Lumbar Spine and total hip bone mineral density | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Toshio Matsumoto, MD, Principal Investigator — Department of Medicine and Bioregulatory Sciences, Universitof Tokushima Graduate School of Health Bioscience

REFERENCES:
- [Derived] Shiraki M, Saito H, Matsumoto T. Eldecalcitol normalizes bone turnover markers regardless of their pre-treatment levels. Curr Med Res Opin. 2012 Sep;28(9):1547-52. doi: 10.1185/03007995.2012.712506. Epub 2012 Aug 23. PMID 22794117
- [Derived] Matsumoto T, Ito M, Hayashi Y, Hirota T, Tanigawara Y, Sone T, Fukunaga M, Shiraki M, Nakamura T. A new active vitamin D3 analog, eldecalcitol, prevents the risk of osteoporotic fractures--a randomized, active comparator, double-blind study. Bone. 2011 Oct;49(4):605-12. doi: 10.1016/j.bone.2011.07.011. Epub 2011 Jul 19. PMID 21784190